CLINICAL TRIAL: NCT03329586
Title: High-intensity Training Safely Improves Exercise Capacity in Heart, Lung, Kidney, and Liver Transplant Recipients
Brief Title: High-intensity Training Safely Improves Exercise Capacity in Heart, Lung, Kidney, and Liver Transplant Recipients: a Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exercise in transplantation
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Physical Activity After Organ Transplantation
Keywords: maximum oxygen consumption; organ transplantation; physical fitness; rehabilitation
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental)
  Interventions: Other: High-intensity training

INTERVENTIONS:
Other: High-intensity training — 6-month individualized home- and group-based training program with the goal to cycle the Mont Ventoux in France

SUMMARY:
The investigators will investigate whether high-intensity exercise training can safely improve physical performance in long-term stable heart, kidney, lung, and liver transplant recipients. Adult transplant recipients will participate in Transplantoux, a 6-month individualized home- and group-based training program, with the goal to cycle the Mont Ventoux in France. The investigators will do cardiopulmonary exercise testing : maximal oxygen consumption, maximal power and BMI.

ELIGIBILITY:
Inclusion Criteria:

* minimum post-transplant period of 6 months
* no acute rejection during the immediately preceding 6 months

Exclusion Criteria:

* patients with cardiovascular or orthopedic contra-indications for intensive physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-06-21 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
VO2max | 6 months after start training
  Maximal oxygen consumption

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Belgium